CLINICAL TRIAL: NCT05475236
Title: Brain Networks of Turning Performance With Aging and Stroke
Brief Title: Neural Underpinnings of Turning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: N3954-M; 1IK1RX003954-01A1 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Aging
Keywords: Aging; Walking; Brain; Transcranial Magnetic Stimulation; Turning

STUDY DESIGN:
Intervention Model Description: Participants will randomized to either receive transcranial direct current stimulation (tDCS) or sham
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told which group (tDCS or sham) they are assigned to. Outcomes Assessors will not be told which group the participant was randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Stimulation (Sham Comparator): Participants will undergo 30 seconds of 2 mA electrical current to the head through saline soaked electrodes.
  Interventions: Behavioral: Experimental: Locomotor Learning
- Transcranial Direct Current Simulation (Experimental): Participants will undergo 20 minutes of 2 mA electrical stimulation to the head through saline soaked electrodes.
  Interventions: Behavioral: Experimental: Locomotor Learning

INTERVENTIONS:
Behavioral: Experimental: Locomotor Learning — Participants will undergo four sessions of locomotor and turn learning. Locomotor learning will involve practicing walking over different terrains (i.e., soft and firm mats) and obstacles at different walking speeds (slow or fast) and turning practice at each end of the walking course. The full cohort will undergo either transcranial direct current stimulation or sham stimulation.

SUMMARY:
Older adults and stroke survivors often have difficulty performing complex walking tasks, due in part to changes in the brain. One task often overlooked is turning, which can lead to injury when performed poorly. The investigators will use non-invasive brain stimulation to assess brain activity and relate those observations to turning performance in older adults and stroke survivors.

DETAILED DESCRIPTION:
This study is associated with an ongoing Clinical Trial (NCT03790657) called the CONTROL Walking Study, which combines locomotor learning and a form of non-invasive electrical brain stimulation call transcranial direct current stimulation (tDCS). The CONTROL Walking Study, randomly places participants into one of two experimental groups (transcranial direct current stimulation or sham stimulation). Following group placement participants complete a 2 week long walking and turning locomotor learning intervention while receiving a group dependent the form of tDCS or sham stimulation.

In leveraging the CONTROL Walking Study infrastructure to further examine the neural control of turning while walking, which is often impaired for older adults and people who have had a stroke. This study will assess neurophysiological brain function using transcranial magnetic stimulation (TMS) which is a form of non-invasive brain stimulation as well as assessing multiple forms of turning performance in older adults. Transcranial magnetic stimulation (TMS) will be used to assess cortical inhibitory neurophysiological function in motor networks of the brain. Importantly, recent work demonstrates significant associations between brain excitatory/inhibitory function and turning performance in older adults, although these results remain largely preliminary.

Therefore, the objective of this proposal is to further elucidate associations between neurophysiological function (measured with TMS) and 360 degree and 180 degree turning performance. The investigators will address the following specific aims:

Specific Aim 1 will test the hypothesis that greater cortical inhibition will be associated with shorter turn duration for 360 degree turns and 180 degree turns.

Specific Aim 2 will test the hypothesis that participants with greater baseline cortical inhibition will demonstrate larger 360 degree and 180 degree turning performance gains (i.e., shorter turn durations).

This new knowledge will provide additional information as to the neural mechanisms associated with turning performance in older adults. Moreover, these results could reveal mechanistic targets for future interventions to enhance turning performance learning and retention.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* preferred 10m walking speed < 1.1 m/s
* self-report of "some difficulty with walking tasks, such as becoming tired when walking a quarter mile, or when climbing two flights of stairs, or when performing household chores."
* Willingness to be randomized to either study group and to participate in all aspects of study assessment and intervention

Exclusion Criteria:

* Diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition (Alzheimer's, Parkinson's, stroke, etc.)
* Contraindications to non-invasive brain stimulation (e.g., metal in head, wound on scalp)
* Contraindications to magnetic resonance imaging (e.g., metal in body, claustrophobia, etc).
* Use of medications affecting the central nervous system
* severe arthritis, such as awaiting joint replacement
* severe obesity (body mass index > 35)
* current cardiovascular, lung or renal disease; diabetes; terminal illness
* myocardial infarction or major heart surgery in the previous year
* cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis (e.g., early stage breast or prostate cancer)
* current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* bone fracture or joint replacement in the previous six months
* current participation in physical therapy for lower extremity function or cardiopulmonary rehabilitation
* current enrollment in any clinical trial
* difficulty communicating with study personnel, and/or non-English speaking
* planning to relocate out of the area during the study period
* clinical judgment of investigative team regarding safety or non-compliance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton W Swanson, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited dataset will be created and shared pursuant to a Data Use Agreement appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, ICF
Time Frame: The Limited Dataset will be completed after the study is completed and primary/secondary data accepted for publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Started | 11 | 5
Completed (This study represents a sub-set of participants from a different clinical trial (NCT03790657). Which investigated the effects of locomotor learning paired with either active or sham tDCS. Only a subset of participants enrolled in NCT03790657 were included, which aimed to further examine the neural control of turning while walking.) | 11 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 11 | 5 | 16
Age, Continuous [Mean (Full Range); unit: years] | 70 [66 to 76] | 72 [65 to 80] | 71.4 [65 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 5 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 5 | 16
Height [Mean (Full Range); unit: Meters (m)] | 1.71 [1.55 to 1.93] | 1.73 [1.63 to 2.00] | 1.73 [1.55 to 2.00]
Weight [Mean (Full Range); unit: Kilograms (kg)] | 83.38 [54.43 to 140.16] | 74.84 [54.43 to 93.89] | 80.71 [54.43 to 140.16]
BMI [Mean (Full Range); unit: weight (kg) / [height (m)]2] | 27.90 [19.97 to 38.41] | 24.74 [19.97 to 32.42] | 26.91 [19.97 to 38.41]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Cortical Silent Period (CSP) (ms)
Description: Cortical Silent Period (CSP) is a single-pulse TMS measure of GABA-mediated cortical inhibition, in which stimulation is applied to the motor cortex while participants are activating a target muscle (here, the tibialis anterior muscle), resulting in a brief reduction in muscle activity. CSP is measured as the time during which the muscle activity is less than the pre-simulation muscle activity level until the return of voluntary muscle activity. CSP is measured in milliseconds (ms).
Time Frame: 30 minutes, Measured at Baseline
Population: Cortical silent period (CSP) data could not be collected from eight participants in the sham group and four participants in the active tDCS group. In these cases, a reliable cortical stimulation site (i.e., motor hotspot) and consistent motor evoked potential (MEP) responses could not be identified, which are required to determine the resting motor threshold necessary for CSP assessment.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Number analyzed (Participants) | 3 | 4
milliseconds (ms) | 104.34 (34.93) | 99.71 (40.45)

2. Primary Outcome: 360 Degree Turn Duration From Baseline
Description: Change in 360 degree turn duration during a 360 degree turn test
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Population: There was a data collection error for one participant in the sham group. There was one data collection error and one participant withdrawal in the tDCS group.
Measure: Mean (Full Range); unit: Seconds (s)
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Number analyzed (Participants) | 10 | 3
Seconds (s) | 0.306 [-0.1 to 0.98] | .367 [0.24 to 0.43]

3. Primary Outcome: 180 Degree Turn Duration From Baseline
Description: Change in 180 degree turn duration as measured during a 2 minute walking task where participants walk back and forth down a corridor.
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Population: One participant from both groups had data collection errors, one additional participant from the active tDCS group withdrew from the study.
Measure: Mean (Full Range); unit: Seconds (s)
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Number analyzed (Participants) | 10 | 3
Seconds (s) | 0.11 [-0.725 to 0.94] | 0.22 [0.04 to 0.49]

4. Primary Outcome: Resting Motor Threshold (Percent of Machine Output)
Description: Resting motor threshold (rMT) is obtained by single-pulse TMS and assesses voltage-gated sodium-channel-mediated cortical excitability. rMT is the minimum intensity (% machine output) of stimulation needed to repeatedly evoke a motor evoked potential (MEP) of at least 50 microvolts in over 50% of trials. It is reported as a percentage of total machine output.
Time Frame: 20 minutes, Measured at Baseline
Population: Reliable cortical stimulation site (i.e., motor hotspot) and consistent motor evoked potential (MEP) responses could not be identified, which are required to determine the resting motor threshold.
Measure: Mean (Full Range); unit: % Maximal Stimulator Output (%MSO)
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Number analyzed (Participants) | 3 | 4
% Maximal Stimulator Output (%MSO) | 56.13 [47.5 to 63.5] | 68.25 [59 to 72]

5. Secondary Outcome: Katz Independence Questionnaire
Description: 6-item participant reported questionnaire assessing level of independence [bathing, dressing, toileting, transferring, continence, feeding]. Total scores range: 0-6, the higher the score, the more independent.
Time Frame: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
Number analyzed (Participants) | 11 | 5
score on a scale | 6 [6 to 6] | 6 [6 to 6]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the baseline visit through the follow-up visit, approximately 3 weeks later (i.e., a monitoring period of about 3 weeks per participant).
Arm/Group | Sham Stimulation | Transcranial Direct Current Simulation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 0/11 | 0/5

LIMITATIONS AND CAVEATS:
Technical challenges during TMS data collection led to incomplete or unreliable neurophysiological data for several participants, limiting the interpretability of outcomes. Additionally, the overall sample size was small, which constrains the generalizability of the findings. The TMS component of the protocol required an FDA risk determination, which delayed the initiation of data collection and further contributed to the limited number of participants available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT05475236/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05475236/ICF_002.pdf